CLINICAL TRIAL: NCT01010776
Title: A Study to Evaluate Switching From Risperidone to Paliperidone ER (Extended Release) in the Treatment of Stable But Symptomatic Schizophrenia Outpatients: Patients Satisfaction and Quality of Life
Brief Title: A Study to Evaluate Participants Satisfaction, Quality of Life and Effectiveness of Flexible-Dose of Paliperidone Extended Release (ER) in Participants With Schizophrenia, Previously Treated With Risperidone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013744; R076477SCH4011 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2009-11-05; First posted 2009-11-10 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental): Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) will be administered orally once daily for 26 weeks of Main Phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
  Interventions: Drug: Paliperidone Extended Release (ER)

INTERVENTIONS:
Drug: Paliperidone Extended Release (ER) — Paliperidone ER tablets in the flexible dose ranging from 3 to 12 mg will be administered orally once daily for 26 weeks of Main Phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.

SUMMARY:
The purpose of this study is to evaluate effectiveness, tolerability (how well a participant can stand a particular medicine or treatment), and safety of flexible-dose of paliperidone extended release (ER) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self), previously taking risperidone (an antipsychotic), but who are not satisfied with their treatment.

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), multi-center (when more than 1 hospital or medical school team work on a medical research study), non-randomized, single-arm study of paliperidone ER in participants previously treated with risperidone with poor response. The study will consist of 2 phases: a main phase of 6 months and an extension phase of another 6 months. The total duration of the study will be 12 months. All participants will receive an oral (having to do with the mouth) daily dose of paliperidone ER in flexible dosage (in the range of 3-12 milligram [mg]: 3 mg, 6 mg, 9 mg, or 12 mg) according to Investigator's discretion. Efficacy and safety of participants will primarily be evaluated by Positive and Negative Syndrome Scale (PANSS) and Extrapyramidal Symptoms Rating Scale (ESRS), respectively. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be postmenopausal (after the time in life when a woman stops having a menstrual period) or surgically sterile or if sexually active, practicing an effective method of birth control (e.g., oral contraceptive, intrauterine device [IUD - an intrauterine device made of plastic and/or copper that is inserted into the womb [uterus] by way of the vaginal canal to used to prevent pregnancy], diaphragm with spermicide [agent that kills spermatozoa] or condom [cover worn over the penis during sexual intercourse to prevent infection or pregnancy] with spermicide) throughout the study and have a negative serum beta - Human Chorionic Gonadotropin (HCG) pregnancy test at screening
* Participants on oral monotherapy (treatment with a single drug) with risperidone in a regimen within the daily dosage recommended by the package insert and adhering to the prescribed risperidone regimen for at least 30 days before entering the study
* Participants with partial response to the current risperidone regimen (persistent symptoms or unstable clinical condition) or presence of unbearable side effects
* Potential Participants switching to another atypical antipsychotic due to their clinical response and/or side effects profile.

Exclusion Criteria:

* Participants with past or current history of psychiatric disease other than schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV
* Participants with concomitant (given at the same time) severe (very serious, life threatening) medical or neurological disorder or risk of suicide
* Participants previously using clozapine
* Participants with a history of previous non-responsiveness to oral antipsychotic treatment
* Pregnant or breast-feeding female participants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (10):
- Brazil (10):
  - Belo Horizonte
  - Criciúma
  - Curitiba
  - Goiânia
  - Itapira
  - Marília
  - Rio de Janeiro
  - Salvador
  - São Paulo
  - Sorocaba

REFERENCES:
- [Derived] Gattaz WF, Campos JA, Lacerda AL, Henna E, Ruschel SI, Bressan RA, de Oliveira IR, Rocha FL, Grabowski HM, Sacomani E Jr, Louza MR, Quevedo J, Elkis H, Zorzetto Filho D, Perico Cde A, Lawson FL, Appolinario JC. Switching from oral risperidone to flexibly dosed oral paliperidone extended-release: core symptoms, satisfaction, and quality of life in patients with stable but symptomatic schizophrenia: the RISPALI study. Curr Med Res Opin. 2014 Apr;30(4):695-709. doi: 10.1185/03007995.2013.869201. Epub 2013 Dec 16. PMID 24289141

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of main phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Period: Main Phase
Arm/Group | Paliperidone Extended Release (ER)
Started | 223
Treated | 218
Completed | 174
Not Completed | 49
Not completed — Withdrawal by Subject | 14
Not completed — Lack of Efficacy | 8
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 6
Not completed — Non-compliance to study medication | 5
Not completed — Selection failure | 2
Not completed — Inform consent withdrawal | 1
Not completed — Other | 1
Not completed — Did not received study medication | 5
Period: In-Between Main Phase & Extension Phase
Arm/Group | Paliperidone Extended Release (ER)
Started | 174
Completed | 159
Not Completed | 15
Not completed — Extension phase was optional | 15
Period: Extension Phase
Arm/Group | Paliperidone Extended Release (ER)
Started | 159
Completed | 156
Not Completed | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone ER - Main Phase Plus Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of main phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER - Main Phase Plus Extension Phase
Number analyzed (Participants) | 218
Age Continuous [Mean (Standard Deviation); unit: Years] | 37.87 (11.01)
Age, Customized [Number; unit: Participants]
  18-21 years | 14
  22-29 years | 50
  30-39 years | 51
  40-49 years | 67
  50-60 years | 35
  61-69 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 139
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 120
  Black | 52
  Oriental | 3
  Mulatto | 9
  Brown | 34
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
  Units on a scale | 94.49 (12.38)
Positive and Negative PANSS Subscales Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS positive subscale assesses 7 positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology). The PANSS negative subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
  Units on a scale
    Positive PANSS Subscale Score | 27.37 (6.48)
    Negative PANSS Subscale Score | 19.76 (5.79)
Personal and Social Performance (PSP) Scale Score [Mean (Standard Deviation); unit: Units on a scale] — The PSP assesses the degree of a participant's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (i, absent to vi, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; =< 30, functioning so poorly as to require intensive supervision.
  Units on a scale | 44.39 (13.11)
Pittsburg Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: Units on a scale] — The PSQI evaluates sleep behavior by means of 7 components: sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disorders, use of sleep medication and daytime dysfunction. The sum of the 7 component scores produces a global score of subjective sleep quality that varies from 0 to 21, with higher scores indicating worse sleep quality.
  Units on a scale | 6.7 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 26 - Main Phase
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Week 26
Population: The intent-to-treat for effectiveness (ITTe) population included all the participants who received at least 1 dose of study medication and provided at least 1 post-baseline effectiveness measurement. Last Observation Carried Forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone Extended Release (ER) - Main Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone Extended Release (ER) - Main Phase
Number analyzed (Participants) | 213
Units on a scale | -22.9 (20.1) [-25.6 to -20.2]

2. Primary Outcome: Change From Baseline in PANSS Total Score at Week 52 - Main Phase Plus Extension Phase
Description: as for outcome 1
Time Frame: Baseline and Week 52
Population: The ITTe population included all the participants who received at least 1 dose of study medication and provided at least 1 post-baseline effectiveness measurement. LOCF method was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone (ER) - Main Phase Plus Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone (ER) - Main Phase Plus Extension Phase
Number analyzed (Participants) | 159
Units on a scale
  Baseline | 93.25 (11.6)
  Change at Week 52 | -26.4 (17.5) [-29.2 to -23.7]

3. Secondary Outcome: Percentage of Participants With Treatment Response in PANSS Total Score - Main Phase
Description: Participants with response in PANSS total score was defined as participants with greater than or equal to 20 percent reduction in PANSS total score from Baseline. The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Paliperidone ER-Main Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER-Main Phase
Number analyzed (Participants) | 213
Percentage of participants | 60.1 [53.2 to 66.7]

4. Secondary Outcome: Percentage of Participants With Treatment Response in PANSS Total Score - Main Phase Plus Extension Phase
Description: as for outcome 3
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Paliperidone ER-Main Phase Plus Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) will be administered orally once daily for 26 weeks of Main Phase. and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER-Main Phase Plus Extension Phase
Number analyzed (Participants) | 159
Percentage of participants | 71.1 [63.4 to 78.0]

5. Secondary Outcome: Change From Baseline in Positive and Negative PANSS Subscales Score at Week 4, 8, 13 and 26 - Main Phase
Description: The PANSS positive subscale assesses 7 positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology). The PANSS negative subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline, Week 4, 8, 13 and 26
Population: The ITTe population included all the participants who received at least 1 dose of study medication and provided at least 1 post-baseline effectiveness measurement. Here 'N' specifies those participants who were evaluated for this outcome measure and 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase
Number analyzed (Participants) | 203
Units on a scale
  Change at Week 4: PANSS positive subscale (n=201) | -3.6 (4.8) [-24.0 to 9.0]
  Change at Week 4: PANSS negative subscale (n=201) | -3.6 (4.8) [-24.0 to 9.0]
  Change at Week 8: PANSS positive subscale (n=191) | -5.0 (5.8) [-25.0 to 20.0]
  Change at Week 8: PANSS negative subscale (n=191) | -5.0 (5.8) [-25.0 to 20.0]
  Change at Week 13: PANSS positive subscale (n=182) | -5.9 (5.8) [-25.0 to 9.0]
  Change at Week 13: PANSS negative subscale (n=182) | -5.9 (5.8) [-25.0 to 9.0]
  Change at Week 26: PANSS positive subscale (n=203) | -5.9 (6.2) [-25.0 to 14.0]
  Change at Week 26: PANSS negative subscale (n=203) | -5.9 (6.2) [-25.0 to 14.0]

6. Secondary Outcome: Change From Baseline in Positive and Negative PANSS Subscales Score at Week 4, 8, 13, 26, 39 and 52 - Main Phase Plus Extension Phase
Description: as for outcome 5
Time Frame: Baseline, Week 4, 8, 13, 26, 39 and 52
Population: The ITTe population included all the participants who received at least 1 dose of study medication and provided at least 1 post-baseline effectiveness measurement. Here 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase Plus Extension Phase
Number analyzed (Participants) | 159
Units on a scale
  Baseline: PANSS positive subscale (n=159) | 26.65 (6.20) [lower limit 6.20]
  Baseline: PANSS negative subscale (n=159) | 19.25 (5.86) [lower limit 5.86]
  Change at Week 4: PANSS positive subscale (n=159) | -3.4 (4.4) [-14.0 to 9.0]
  Change at Week 4: PANSS negative subscale (n=159) | -3.4 (4.4) [-14.0 to 9.0]
  Change at Week 8: PANSS positive subscale (n=159) | -5.4 (5.1) [-18.0 to 9.0]
  Change at Week 8: PANSS negative subscale (n=159) | -5.4 (5.1) [-18.0 to 9.0]
  Change at Week 13: PANSS positive subscale (n=159) | -5.9 (5.7) [-18.0 to 9.0]
  Change at Week 13: PANSS negative subscale (n=159) | -5.9 (5.7) [-18.0 to 9.0]
  Change at Week 26: PANSS positive subscale (n=159) | -6.8 (5.5) [-20.0 to 9.0]
  Change at Week 26: PANSS negative subscale (n=159) | -6.8 (5.5) [-20.0 to 9.0]
  Change at Week 39: PANSS positive subcale (n=152) | -7.3 (5.9) [-25.0 to 4.0]
  Change at Week 39: PANSS negative subscale (n=152) | -7.3 (5.9) [-25.0 to 4.0]
  Change at Week 52: PANSS positive subscale (n=154) | -7.5 (6.1) [-25.0 to 10.0]
  Change at Week 52: PANSS negative subscale (n=154) | -7.5 (6.1) [-25.0 to 10.0]

7. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Scale Score at Week 4, 8, 13 and 26 - Main Phase
Description: The PSP scale evaluates the dysfunction degree exhibited by the participants, regarding 4 behavioral domains: useful social activities, personal and social relations, self-care and agitated and aggressive behavior. Each domain were assessed on a 6-point scale (0=absent to 5=very severe). A transformed score from 1 to 100 is generated from the raw score based on the clinical interpretation of the scores generated in the 4 areas of functioning, with a higher transformed score indicating better function.
Time Frame: Baseline, Week 4, 8, 13 and 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase
Number analyzed (Participants) | 204
Units on a scale
  Change at Week 4 (n=201) | 5.7 (11.7)
  Change at Week 8 (n=191) | 8.3 (12.8)
  Change at Week 13 (n=182) | 9.9 (14.8)
  Change at Week 26 (n=204) | 10.4 (14.9)

8. Secondary Outcome: Change From Baseline in PSP Scale Score at Week 4, 8, 13, 26, 39 and 52 - Main Phase Plus Extension Phase
Description: as for outcome 7
Time Frame: Baseline, Week 4, 8, 13, 26, 39 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase Plus Extension Phase
Number analyzed (Participants) | 159
Units on a scale
  Baseline (n=159) | 45.17 (12.84)
  Change at Week 4 (n=159) | 5.3 (9.6)
  Change at Week 8 (n=159) | 9.0 (12.6)
  Change at Week 13 (n=159) | 9.7 (14.4)
  Change at Week 26 (n=159) | 12.0 (12.7)
  Change at Week 39 (n=151) | 12.6 (14.2)
  Change at Week 52 (n=155) | 14.6 (14.9)

9. Secondary Outcome: Change From Baseline in Pittsburg Sleep Quality Index (PSQI) Score at Week 4, 8, 13 and 26 - Main Phase
Description: The PSQI evaluates sleep behavior by means of 7 components: sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disorders, use of sleep medication and daytime dysfunction. The sum of the 7 component scores produces a global score of subjective sleep quality that varies from 0 to 21, with higher scores indicating worse sleep quality.
Time Frame: Baseline, Week 4, 8, 13 and 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase
Number analyzed (Participants) | 198
Units on a scale
  Baseline (n=198) | 6.7 (4.1)
  Change at Week 4 (n=174) | -1.0 (3.5)
  Change at Week 8 (n=162) | -1.2 (3.5)
  Change at Week 13 (n=156) | -1.5 (3.3)
  Change at Week 26 (n=174) | -1.4 (3.7)

10. Secondary Outcome: Change From Baseline PSQI Score at Week 4, 8, 13, 26, 39 and 52 - Main Phase Plus Extension Phase
Description: as for outcome 9
Time Frame: Baseline, Week 4, 8, 13, 26, 39 and 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase Plus Extension Phase
Number analyzed (Participants) | 148
Units on a scale
  Baseline (n=148) | 6.4 (4.1)
  Change at Week 4 (n=140) | -1.0 (3.6)
  Change at Week 8 (n=136) | -1.3 (3.2)
  Change at Week 13 (137) | -1.5 (3.2)
  Change at Week 26 (n=135) | -1.4 (3.5)
  Change at Week 39 (n=133) | -1.9 (3.9)
  Change at Week 52 (n=133) | -1.9 (3.4)

11. Secondary Outcome: Number of Participants With Clinical Global Impression-Severity (CGI-S) Score - Main Phase
Description: The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant.The categories included in the scale are normal, without any disease, borderline, slightly ill, moderately ill, markedly ill, severely ill and extremely ill. A rating of 1="Normal, not at all ill" and a rating of 7 ="Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, Week 4, 8, 13 and 26
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Paliperidone ER-Main Phase
Number analyzed (Participants) | 213
Participants
  Baseline: Borderline (n=213) | 2
  Baseline: Slightly ill (n=213) | 4
  Baseline: Moderately ill (n=213) | 52
  Baseline: Markedly ill (n=213) | 114
  Baseline: Severely ill (n=213) | 40
  Baseline: Extremely ill (n=213) | 1
  Week 4: Borderline (n=201) | 4
  Week 4: Slightly ill (n=201) | 25
  Week 4: Moderately ill (n=201) | 87
  Week 4: Markedly ill (n=201) | 61
  Week 4: Severely ill (n=201) | 24
  Week 8: Borderline (n=191) | 5
  Week 8: Slightly ill (n=191) | 35
  Week 8: Moderately ill (n=191) | 80
  Week 8: Markedly ill (n=191) | 56
  Week 8: Severely ill (n=191) | 15
  Week 8: extremely ill (n=191) | 0
  Week 13: Normal, without any disease (n=182) | 2
  Week 13: Borderline (n=182) | 7
  Week 13: Slightly ill (n=182) | 41
  Week 13: Moderately ill (n=182) | 73
  Week 13: Markedly ill (n=182) | 47
  Week 13: Severly ill (n=182) | 12
  Week 26: Normal without any disease (n=204) | 3
  Week 26: Borderline (n=204) | 16
  Week 26: Slightly ill (n=204) | 48
  Week 26: Moderately ill (n=204) | 70
  Week 26: Markedely ill (n=204) | 48
  Week 26: Severely ill (n=204) | 19

12. Secondary Outcome: Number of Participants With Clinical Global Impression-Severity (CGI-S) Score - Extension Phase
Description: as for outcome 11
Time Frame: Week 39 and 52
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- Paliperidone ER - Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally, once daily for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER - Extension Phase
Number analyzed (Participants) | 155
Participants
  Week 39: Normal without any disease (n=152) | 2
  Week 39: Borderline (n=152) | 22
  Week 39: Slightly ill (n=152) | 41
  Week 39: Moderately ill (n=152) | 55
  Week 39: Markedely ill (n=152) | 22
  Week 39: Severely ill (n=152) | 10
  Week 52: Borderline (n=155) | 23
  Week 52: Slightly ill (n=155) | 37
  Week 52: Moderately ill (n=155) | 58
  Week 52: Markedely ill (n=155) | 24
  Week 52: Severely ill (n=155) | 10

13. Secondary Outcome: Percentage of Participants With Treatment Satisfaction - Main Phase
Description: Participant's response regarding satisfaction with the treatment were recorded. A 5-point evaluation scale was used to evaluate participant satisfaction: very good, good, moderate, bad and very bad.
Time Frame: Baseline, Week 4, 8, 13 and 26
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Groups:
- Paliperidone ER - Main Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER - Main Phase
Number analyzed (Participants) | 213
Percentage of Participants
  Baseline: Very good (n=213) | 11.7
  Baseline: Good (n=213) | 38.5
  Baseline: Moderate (n=213) | 34.3
  Baseline: Bad (n=213) | 12.7
  Baseline: Very bad (n=213) | 2.8
  Week 4: Very good (n=200) | 29.5
  Week 4: Good (n=200) | 52.5
  Week 4: Moderate (n=200) | 16.5
  Week 4: Bad (n=200) | 1.0
  Week 4: Very bad (n=200) | 0.5
  Week 8: Very good (n=190) | 33.7
  Week 8: Good (n=190) | 48.9
  Week 8: Moderate (n=190) | 13.7
  Week 8: Bad (n=190) | 3.7
  Week 13: Very good (n=182) | 37.4
  Week 13: Good (n=182) | 46.2
  Week 13: Moderate (n=182) | 12.1
  Week 13: Bad (n=182) | 3.8
  Week 13: Very bad (n=182) | 0.5
  Week 26: Very good (n=204) | 36.3
  Week 26: Good (n=204) | 46.1
  Week 26: Moderate (n=204) | 10.8
  Week 26: Bad (n=204) | 4.4
  Week 26: Very bad (n=204) | 2.5

14. Secondary Outcome: Percentage of Participants With Treatment Satisfaction-Main Phase Plus Extension Phase
Description: as for outcome 13
Time Frame: Baseline, Week 4, 8, 13, 26, 39 and 52
Population: The ITTe population included all the participants who received at least 1 dose of study medication and provided at least 1 post-baseline effectiveness measurement. 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Number; unit: Percentage of participants
Groups:
- Paliperidone ER-Main Phase Plus Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER-Main Phase Plus Extension Phase
Number analyzed (Participants) | 159
Percentage of participants
  Baseline: Very good (n=159) | 13.2
  Baseline: Good (n=159) | 40.9
  Baseline: Moderate (n=159) | 32.1
  Baseline: Bad (n=159) | 11.3
  Baseline: Very bad (n=159) | 2.5
  Week 4: Very good (n=159) | 31.4
  Week 4: Good (n=159) | 54.1
  Week 4: Moderate (n=159) | 13.8
  Week 4: Very bad (n=159) | 0.6
  Week 8: Very good (n=159) | 37.1
  Week 8: Moderate (n=159) | 11.3
  Week 8: Bad (n=159) | 3.1
  Week 13: Very good (n=159) | 39.0
  Week 13: Good (n=159) | 46.5
  Week 13: Moderate (n=159) | 10.1
  Week 13: Bad (n=159) | 3.8
  Week 13: Very bad (n=159) | 0.6
  Week 26: Very good (n=159) | 41.5
  Week 26: Good (n=159) | 50.9
  Week 26: Moderate (n=159) | 6.9
  Week 26: Very bad (n=159) | 0.6
  Week 39: Very good (n=152) | 38.8
  Week 39: Good (n=152) | 51.3
  Week 39: Moderate (n=152) | 7.2
  Week 39: Bad (n=152) | 2.0
  Week 39: Very bad (n=152) | 0.7
  Week 52: Very good (n=155) | 41.3
  Week 52: Good (n=155) | 43.2
  Week 52: Moderate (n=155) | 12.9
  Week 52: Bad (n=155) | 2.6

15. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) Score - Main Phase
Description: The SF-36 is designed to assess the health status of participants. The SF-36 includes 1 multi-item scale measuring physical health component and mental health component. Physical health component includes physical functioning, role limitations due to physical health, pain and general health. Mental health component includes role limitations due to emotional problems, energy/fatigue, emotional well being and social functioning. Each item is scored on a 0-100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state. The score for a component (physical or mental) is an average of the individual item scores. Each component is scored on a scale of 1 to 100, where 100=highest level of functioning.
Time Frame: Baseline and Week 26
Population: The ITTe population included all the participants who received at least 1 dose of study medication and provided at least 1 post-baseline effectiveness measurement. Here 'N' specifies those participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone ER- Main Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER- Main Phase
Number analyzed (Participants) | 190
Units on a scale
  Baseline: Physical component summary | 47.9 (8.8)
  Baseline: Mental component summary | 35.9 (8.5)
  Week 26: Physical component summary | 48.4 (7.6)
  Week 26: Mental component summary | 38.3 (8.0)

16. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) Score - Main Phase Plus Extension Phase
Description: as for outcome 15
Time Frame: Baseline and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone ER-Main Phase Plus Extension Phase
Number analyzed (Participants) | 150
Units on a scale
  Baseline: Physical component summary | 48.7 (8.6)
  Baseline: Mental component summary | 35.7 (8.5)
  Week 52: Physical component summary | 48.8 (7.6)
  Week 52: Mental component summary | 38.5 (8.4)

17. Other Pre Specified Outcome: Change From Baseline in Extrapyradimal Symptoms Rating Scale (ESRS) Total Score at Week 4, 8, 13 and 26 - Main Phase
Description: An ESRS scale is used to assess the extrapyramidal symptoms attributable to antipsychotics. It consists of 8 items to assess individual symptoms and each item is assessed from 0 (none, normal) to 4 (severe). The total score is the sum of the 8 item scores, for a total range of 0 (normal) to 32 (severe). The items for the assessment of individual symptoms are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia.
Time Frame: Baseline, Week 4, 8, 13 and 26
Population: The safety analysis population included all the participants that received at least one dose of study medication and provided any post-baseline information. Here 'N' specifies those participants who were evaluated for this outcome measure and 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone ER - Main Phase: Single oral dose of paliperidone ER tablet within the range of 3 to 12 mg once a day was administered for 26 weeks. Dosage was adjusted as per the investigator's discretion.
Arm/Group | Paliperidone ER - Main Phase
Number analyzed (Participants) | 215
Units on a scale
  Baseline (n=215) | 1.30 (1.99)
  Change at Week 4 (n=201) | -0.40 (1.23)
  Change at Week 8 (n=189) | -0.45 (1.47)
  Change at Week 13 (n=182) | -0.63 (1.76)
  Change at Week 26 (n=201) | -0.6 (1.71)

18. Other Pre Specified Outcome: Change From Baseline in ESRS Total Score at Week 4, 8, 13, 26, 39 and 52 - Main Phase Plus Extension Phase
Description: as for outcome 17
Time Frame: Baseline, Week 4, 8, 13, 26, 39 and 52
Population: The safety analysis population included all the participants that received at least 1 dose of study medication and provided 1 post-baseline information. Here 'N' specifies those participants who were evaluated for this outcome measure and 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone ER-Main Plus Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER-Main Plus Extension Phase
Number analyzed (Participants) | 159
Units on a scale
  Baseline (n=159) | 1.41 (2.14)
  Change at Week 4 (n=159) | -0.51 (1.31)
  Change at Week 8 (n=159) | -0.49 (1.56)
  Change at Week 13 (n=159) | -0.68 (1.85)
  Change at Week 26 (n=158) | -0.77 (1.87)
  Change at Week 39 (n=151) | -0.81 (1.97)
  Change at Week 52 (n=154) | -0.75 (1.94)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: The safety analysis population included all the participants that received at least 1 dose of study medication and provided 1 post-baseline information. Here, 215 and 159 participants were inculded in safety analysis set for main phase and extension phase, respectively.
Groups:
- Paliperidone ER - Extension Phase: Paliperidone ER tablets in the flexible dose ranging from 3 to 12 milligram (mg) was administered orally once daily for 26 weeks of Main Phase and for additional 26 weeks of Extension Phase to participants who continued with Extension Phase. Dosage was adjusted as per the Investigator's discretion.
Arm/Group | Paliperidone ER - Main Phase | Paliperidone ER - Extension Phase
Serious Adverse Events (participants affected / at risk) | 14/215 | 3/159
Other Adverse Events (participants affected / at risk) | 144/215 | 70/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER - Main Phase (N=215) | Paliperidone ER - Extension Phase (N=159)
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Psychomotor agitation (Psychiatric disorders) | 1 | 0
Psychotic disorder NOS (Psychiatric disorders) | 5 | 0
Schizophrenia NOS (Psychiatric disorders) | 2 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Hospitalization (Surgical and medical procedures) | 2 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Pregnancy NOS (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER - Main Phase (N=215) | Paliperidone ER - Extension Phase (N=159)
Insomnia (Psychiatric disorders) | 32 | 14
Anxiety (Psychiatric disorders) | 23 | 4
Depression (Psychiatric disorders) | 8 | 7
Agitation (Psychiatric disorders) | 12 | 0
Psychotic disorder NOS (Psychiatric disorders) | 7 | 0
Libido decreased (Psychiatric disorders) | 3 | 2
Schizophrenia NOS (Psychiatric disorders) | 4 | 0
Psychomotor retardation (Psychiatric disorders) | 2 | 1
Nervousness (Psychiatric disorders) | 2 | 1
Aggression (Psychiatric disorders) | 2 | 1
Logorrhea (Psychiatric disorders) | 2 | 0
Obsessive thoughts (Psychiatric disorders) | 1 | 1
Impulsive behavior NOS (Psychiatric disorders) | 1 | 1
Hostility (Psychiatric disorders) | 1 | 1
Hallucination NOS (Psychiatric disorders) | 2 | 0
Depressive symptom (Psychiatric disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Sleep disorder NOS (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Psychomotor agitation (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Somnolence (Nervous system disorders) | 13 | 4
Headache (Nervous system disorders) | 13 | 4
Akathisia (Nervous system disorders) | 8 | 5
Psychomotor hyperactivity (Nervous system disorders) | 8 | 0
Tremor (Nervous system disorders) | 6 | 0
Parkinsonism (Nervous system disorders) | 6 | 0
Dizziness (Nervous system disorders) | 6 | 0
Dystonia (Nervous system disorders) | 4 | 0
Extrapyramidal disorder (Nervous system disorders) | 2 | 1
Sedation (Nervous system disorders) | 3 | 0
Aphonia (Nervous system disorders) | 1 | 1
Ageusia (Nervous system disorders) | 1 | 1
Speech disorder (Nervous system disorders) | 2 | 0
Hypokinesia (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Repetitive speech (Nervous system disorders) | 1 | 0
Weight increased (Investigations) | 23 | 20
Weight decreased (Investigations) | 5 | 5
Blood triglycerides increased (Investigations) | 2 | 2
Blood prolactin increased (Investigations) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Vomiting NOS (Gastrointestinal disorders) | 2 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Gastritis NOS (Gastrointestinal disorders) | 0 | 1
Food poisoning NOS (Gastrointestinal disorders) | 1 | 0
Aptyalism (Gastrointestinal disorders) | 1 | 0
Dyslipidemia (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus NOS (Metabolism and nutrition disorders) | 2 | 2
Appetite decreased NOS (Metabolism and nutrition disorders) | 3 | 0
Appetite increased NOS (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Malaise (General disorders) | 3 | 0
Pain NOS (General disorders) | 1 | 1
Influenza like illness (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 1
Feeling abnormal (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Erectile dysfunction NOS (Reproductive system and breast disorders) | 2 | 2
Ejaculation failure (Reproductive system and breast disorders) | 1 | 1
Breast discharge (Reproductive system and breast disorders) | 0 | 1
Hypertension NOS (Vascular disorders) | 4 | 3
Hypertensive crisis (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Infected sebaceous cyst (Infections and infestations) | 1 | 0
Sinusitis NOS (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Skin lesion NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Acne NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hospitalization (Surgical and medical procedures) | 3 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Eye movement disorder NOS (Eye disorders) | 1 | 0
Tachycardia NOS (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypersensitivity NOS (Immune system disorders) | 1 | 0
Lower limb fracture NOS (Injury, poisoning and procedural complications) | 1 | 0
Mycosis fungoides NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Galactorrhea (Reproductive system and breast disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The Sponsor can require changes to the communication and can extend the embargo.